CLINICAL TRIAL: NCT03921385
Title: Augmented Reality Enhanced Surgery: Proof-of-concept Study for the Use of Holographic Technology in Cranial and Spinal Surgery
Brief Title: Augmented Reality Enhanced Surgery: Use of Holographic Technology in Cranial and Spinal Surgery
Acronym: ARinOR
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 828346
Record Dates: First submitted 2018-02-23; First posted 2019-04-19 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single cohort - navigated cranial and spine surgery
  Interventions: Device: Augmented Reality Headset

INTERVENTIONS:
Device: Augmented Reality Headset — Patients undergoing navigated cranial or spine procedures will acquire standard of care clinical high-resolution imaging to be used for registration purposes intraoperatively. VGA output on the navigation machine will be utilized to project imaging information to the augmented reality headset. The holographic image will then be recorded to assess feasibility and ease of use.

SUMMARY:
* To demonstrate the feasibility of integrating holographic technology as a heads-up display for navigated cranial and spinal neurosurgical procedures. This entails simply displaying the navigation screen currently used by Medtronic Stealth or Brainlab systems as a holographic image that can be positioned closer to the operative field.
* To develop a systematic, efficient communication and registration process allowing holographic technology to be potentially utilized as a navigation tool in cranial and spinal neurosurgery. This entails developing software, optimizing connection parameters, and devising registration techniques incorporating line-of-sight fiducial markers to allow the holographic device to function as a navigation instrument.

ELIGIBILITY:
Inclusion Criteria:

* age >= 18
* must be able to read and understand English, and sign the informed consent form

Exclusion Criteria:

* emergent/emergency procedures
* pediatric patients
* pregnant patients
* vulnerable populations

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Any patient undergoing an elective cranial or spinal procedure at the University of Pennsylvania, Department of Neurosurgery.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2018-02-22 (Actual); Primary Completion 2019-01-18 (Actual); Study Completion 2022-07-14 (Actual)

PRIMARY OUTCOMES:
Assessment of holographic technology in the operating room using a feasibility scale ranging from 1-10 | 2 years
  To demonstrate the feasibility of integrating holographic technology as a heads-up display for navigated cranial and spinal neurosurgical procedures. This entails simply displaying the navigation screen currently used by Medtronic Stealth or Brainlab systems as a holographic image that can be positioned closer to the operative field.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania Medical Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No